CLINICAL TRIAL: NCT04007042
Title: Validation of a Short Questionnaire (SSI) for Sleep Disorders in Patients With Alcohol
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 12 05 04
Record Dates: First submitted 2019-06-27; First posted 2019-07-05 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Alcohol Dependence; Sleep Disorder
MeSH Terms: conditions — Alcoholism; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sleep disorders are very common in alcohol patients (40-90% according to studies) These sleep disorders may persist after withdrawal and represent a major factor in relapse.

In a previous study, the investigators validated a simple sleep questionnaire (the "Short Sleep Index = SSI") from a multicentre series of 602 American patients (Perney et al., Alcohol Alcohol 2012) The SSI is obtained from the Hamilton score (baseline score for anxiety and depression)

DETAILED DESCRIPTION:
to compare the SSI with a reference sleep questionnaire (Pittsburg Quality Sleep Index) in alcohol patients in different situations: Ambulatory or hospitalization

ELIGIBILITY:
Inclusion Criteria Sick people with alcohol abuse or dependence Inpatient or outpatient follow-up (Nîmes University Hospital, Grau du Roi Hospital, Montpellier, Centre de Soins d'Accompagnement et de Prévention en Addictologie (CSAPA of Nîmes University Hospital) Agreeing to answer the questionnaire Not having a cognitive deficit or psychiatric pathology that makes interrogation unreliable

* Exclusion criteria : NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with alcohol abuse or dependence
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-01-15 (Actual); Primary Completion 2013-01-15 (Actual); Study Completion 2013-01-15 (Actual)

PRIMARY OUTCOMES:
to compare the SSI with a reference sleep questionnaire (Pittsburg Quality Sleep Index | Day 1
  PQSI and SSI scores. PQSI : The overall score is obtained by summing the seven components. It goes from 0: "no difficulty" to 21: "major difficulties".
  A PSQI greater than 5 indicates sleep disturbances and ranks subjects as good and bad sleepers.

SECONDARY OUTCOMES:
compare the duration of these 2 tests | Day 1
  duration (minutes, seconds)